CLINICAL TRIAL: NCT01314196
Title: The Influence of Resistance Training Biceps as an Adjunct to Rehabilitation of the Shoulder in Subacromial Impingement Syndrome (SIS)
Brief Title: Progressive Resistance Training of the Biceps in Subacromial Impingement Syndrome
Acronym: PRTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Jamil Natour, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNCISAL/1019
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2010-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: biceps; resistance training; rehabilitation; impact syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- therapeutic exercises (Active Comparator): therapeutic exercises for the shoulder and scapula stabilizers
  Interventions: Other: therapeutic exercises
- progressive resistance training biceps (Experimental): therapeutic exercises for the shoulder and scapula stabilizers and biceps resistance training.
  Interventions: Other: biceps resistance training and therapeutic exercises

INTERVENTIONS:
Other: therapeutic exercises — therapeutic exercises for the shoulder and scapula stabilizers using bat without charge, training and isometric exercises commuting to the cuff muscles, without producing subacromial impaction.
  Arms: therapeutic exercises
Other: biceps resistance training and therapeutic exercises — The biceps resistance training based on calculations of maximum resistance (MR), being conduct in three series 10 reps with 50% of MR in the first series of training and 75% of MR in the second series, with 2 minutes between each and therapeutic exercises for the shoulder and scapula stabilizers.
  Other Names: progressive resistance training
  Arms: progressive resistance training biceps

SUMMARY:
The aim of this study was to evaluate the influence of progressive resistance training of the biceps in shoulder rehabilitation in patients with subacromial impingement syndrome (SIS).

Method: a randomized controlled clinical trial, with analysis intention-to-treat, approved by the Ethics and Research (1019/08), containing sixty patients of both sexes, SIS, evaluated at the initial time (T0), with 45 days (T45) and 90 days of treatment (T90). We analyzed the pain at rest (VAS), range of shoulder movement, strength, function by The Disabilities of Arm, Shoulder and Hand (DASH) and quality of life by Short Form-36 (SF-36) and Western Ontario Rotator Cuff Index (WORC). They recommended the use of NSAIDs and analgesics in the presence of pain exacerbated, every eight hours. Study groups will perform therapeutic exercises for the shoulder and scapula stabilizers. In the experimental group associate progressive resistance training of the biceps.

DETAILED DESCRIPTION:
Sixty patients in the Physical Therapy Clinic at the University of Health Sciences of Alagoas, of both sexes with a clinical diagnosis of SIS, according to the criteria of Neer. Included will be those with a diagnosis of injury to one or more rotator cuff tendons, with pain for three months or more, ranging from 3 to 8, based on visual analogic scale(VAS) ranging from 0 to 10. Hawkins' test and Neer positive and aged between 18 and 65. The presence of total rupture of the long head of biceps, and associated rheumatic shoulder surgery represented exclusion criteria. After approval by the IRB (1019/08) were prepared sealed envelopes, to maintain the secrecy of allocation, and the patients were divided into control and experimental group and evaluated by a blind assessor, at the initial time (T0), after 45 days of treatment (T45) and 90 days of treatment (T90). The shoulder will be assessed in the degree of active motion for flexion, extension, medial and lateral rotation and abduction, with the patient in standing position using manual goniometer. To determine the movement of flexion and extension, the upper limb was positioned in the sagittal plane, goniometer along the mid-axillary line of the trunk and the axle in the humeral head. The movable arm of the goniometer was placed over the body surface of the humerus toward the lateral epicondyle. Abduction to the fixed arm of the goniometer was positioned over the posterior axillary line of the trunk, aligned with the blade and the moving arm was placed on the posterior surface of the arm along the longitudinal axis of the humerus. The medial and lateral rotation was accomplished by positioning the shoulder in abduction of 90 degrees, the axle of the goniometer positioned on the olecranon and the movable arm along the axis of the forearm.

The strength of manual pressure was assessed using the hydraulic dynamometer, manufactured in Korea. The instrument is graduated in two scales - kilogram force (Maximum 90 pounds), form-fitting and catcher with five adjustment positions to accommodate any size hand during the evaluation. During the strength assessment, the upper limb was positioned at rest beside the body with elbow flexed 90 degrees, forearm and wrist in neutral position.

Pain assessment will be conducted at rest, using VAS ranging from 0 (no pain) to 10 cm (intolerable pain). The Disabilities of The Arm, Shoulder and Hand (DASH) questionnaire was used for the evaluation of impairment and physical symptoms of upper limbs. It consists of 30 mandatory items related to function and symptoms (DASH 1) and two optional areas, divided into four issues for work activities (DASH 2) and 4 questions for activities of daily living (DASH 3). The Western Ontario Rotator Cuff Index (WORC) and Short- form health survey (SF-36) were the tools used to evaluate the quality of life. The WORC is specific to patients suffering from rotator cuff injury with five domains: physical symptoms (SF), sports and recreation (ER), work (T), state of vitality (EV) and emotion (E). The WORC scores can be set by calculation or by the general analysis of independent domains.

The treatment plan will be held for 3 months, twice a week throughout the sample, through the practice of therapeutic exercises for the shoulder and scapula stabilizers using bat without charge, training and isometric exercises commuting to the cuff muscles, without subacromial generate impaction. In the experimental group, we associate the progressive resistance training of the biceps. The progression of resistance training biceps, based on calculations of maximum resistance (MR), being conducted in three sets of 10 repetitions with 50% of MRI in the first series of training and 75% of MRI in the second series, 2 minutes, between each. In the presence of pain greater than or equal to seven, based on the VAS, patients were instructed in the use of paracetamol 750mg every six hours and diclofenac sodium 50mg every eight hours.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical diagnosis of injury to one or more muscles of the rotator cuff;
* pain for three months or more, and pain between three and eight, according to visual analog scale (VAS);
* Hawkins and Neer test positive;
* aged between 18 and 65

Exclusion Criteria:

* fractures of the upper phase of consolidation;
* patients with total rupture of the long head of the biceps due to the impossibility of getting the muscle resistance training;
* patients undergoing surgical procedures for shoulder in the three months preceding the study;
* associated rheumatic diseases because they may interfere in the evaluation of patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain at rest and quality of life | initial time, 45 days and 90 days of treatment
  Pain assessment will be conducted at rest, using VAS ranging from 0 (no pain) to 10 cm (unbearable pain). The Westein Ontario Rotator Cuff Index (WORC) and Short form-36(SF-36) were the instruments used to assess the quality of life.

SECONDARY OUTCOMES:
Evaluation range of motion,strength and physical symptoms of the shoulder | initial time, 45 days and 90 days of treatment
  The range of motion the shoulder will be assessed by goniometry for flexion, extension, medial and lateral rotation and abduction. The strength of manual pressure was assessed using the hydraulic dynamometer, Jamar type, manufactured by Saehan Corporation in Korea. O Disabilities Of The Arm, Shoulder and Hand (DASH), was intended for assessment of physical symptoms and disorders of the upper limbs.

CONTACTS AND LOCATIONS:
Overall Officials: ANA C COÊLHO, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil